CLINICAL TRIAL: NCT03432429
Title: Rapid Evaporative Ionisation Mass Spectrometry for Examination of Circumferential Surgical Excision Margins
Brief Title: Real Time Tissue Characterisation Using Mass Spectrometry REI-EXCISE iKnife Study
Acronym: REI-EXCISE
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Cancer Research UK (Other); Waters Corporation (Unknown)
Responsible Party: Sponsor
Other Study IDs: 13SM1815; 14/EE/0024 (Sub) (Other: REC)
Record Dates: First submitted 2017-11-17; First posted 2018-02-14 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Breast Cancer; Surgery
Keywords: Tumours; Breast conserving surgery; Margin assessment technology; Mass spectrometry
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Resected tissue samples will undergo detailed histopathological examination using a standard reporting schema based on the Royal College of Pathologists guidelines for breast specimen processing and the results of the histological examination of the tissue along the electrosurgical dissection line will be compared to the results of mass spectrometric tissue identification.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: REIMS iKnife — Use of REIMS iKnife in breast conserving surgery

SUMMARY:
REI-EXCISE is a multicentre, prospective, non-randomised feasibility study, aimed to evaluate the diagnostic accuracy of rapid ionisation mass spectroscopy using an iKnife device. The iKnife will collect vapour, a by-product of surgery, which will pass through the mass spectrometer machine for analysis in order to evaluate what is "normal" and what is "cancerous" breast tissue.

DETAILED DESCRIPTION:
There is an urgent need to address high rates of close or positive margins and re-operative breast cancer surgery, which commonly results from the inability of the surgeon to rapidly and reliably evaluate resection margin status intra-operatively.

This study therefore seeks to address this problem by aiming to develop a method for near real time, in vivo intra-operative tissue classification that may be used by breast surgeons as an intelligent knife (or "iKnife") to better guide oncological margin control. The method known as Rapid Evaporative Ionisation Mass Spectrometry (REIMS) technology uses mass spectrometric and chemometric analysis of the tissue specific ionic content of the surgical diathermy smoke plume for the rapid identification of dissected breast tissues.

There are no additional treatment interventions as part of REI-EXCISE. The main study procedures are breast conserving surgery using the REIMS iKnife for mass spectral analysis of each surgical margin and correlation between the results of a software recognition algorithm that capitalised on the spectral data (i.e. iKnife margin = positive / negative) with conventional histopathological assessment. False positive iKnife data will be further interrogated with digital droplet polymerase chain reaction and imprint cytology assessment.

ELIGIBILITY:
Inclusion Criteria:

* BCS for ductal carcinoma in situ (B5a)
* BCS for invasive ductal carcinoma (B5b)
* BCS for invasive lobular carcinoma (B5b)
* B3 lesions undergoing surgical excision

Exclusion Criteria:

* Pregnant or lactating
* 18 years or younger
* Diagnostic excision biopsy for classical lobular carcinoma in situ (LCIS) (current practice is that classical LCIS at a surgical resection margin would not mandate wider excision)

Or if the patient is diagnosed with

• Non-epithelial breast tumour (phyllodes, lymphoma)

Note on patients receiving Neo-adjuvant Chemotherapy (NACT):

Patients selecting to receive NACT will be eligible for participation. However, the data for patients receiving NACT will be analysed separately as a pre-planned subgroup and these patients will not contribute data to the n=35 patients with positive margins required for this feasibility trial. Data from NACT cases have not been used to generate the validated multispectral database since eccentric fibrosis made the histological analysis more complex, which limited the number of patients in whom tissue was available for research.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients undergoing breast conserving surgery (BCS) for invasive or non-invasive breast cancer.
  There is no upper age limit. We believe that older adults represent a group for whom multiple operations could represent a significant perioperative risk and therefore might stand to benefit from iKnife as much if not more so than younger patients. The lower age limit is 18 for the purposes of adequate informed consent to take part in this trial. A breast cancer diagnosis in adolescence is extremely rare.
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2021-12-08 (Actual); Study Completion 2021-12-08 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy | Data collected during recruitment period: 1st June 2017 until 31st May 2019 i.e. 24 months.
  The diagnostic accuracy of rapid ionisation mass spectroscopy for oncological margin status will be measured during breast conserving surgery (BCS) (n=35 patients with positive margins). The primary end-point will allow to report accuracy (sensitivity and specify) of rapid ionisation mass spectroscopy to distinguish between patients with at least one close or positive margin and those without close or positive margin.

SECONDARY OUTCOMES:
Assessment of procedure duration using REIMS | Data collected during recruitment period: 1st June 2017 until 31st May 2019 i.e. 24 months.
  This study will quantify whether REIMS adds significantly to the intra-operative time taken to perform breast conserving surgery. Thus, the data generated with REI-EXCISE trial will report the difference in specimen excision time using iKnife as compared to conventional electrosurgery.
REIMS technology user satisfaction | Data collected during recruitment period: 1st June 2017 until 31st May 2019 i.e. 24 months.
  This study will be collecting data to understand if end-users are sufficiently satisfied with REIMS technology framework (including modified hand-piece) , and are willing to use it routinely during breast conserving surgery (BCS). This will be conveyed by analysing the end user questionnaire completed by the surgeons to infer if they are satisfied with the use of REIMS instrumentation in vivo to perform BCS.
Accuracy of predicting oncological status | Data collected during recruitment period: 1st June 2017 until 31st May 2019 i.e. 24 months.
  The intra-operative REIMS analysis will be used to accurately predict/measure the oncological status of the surface of the wide local excision cavity. The data will be reported as the proportion of patients with all close or positive margins correctly detected as positive by iKnife and as the proportion of patients with no margin malignancy correctly detected by iKnife among the true negative patients.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Leff, Principal Investigator — Department of Surgery & Cancer, Imperial College London; Zoltan Takats, Principal Investigator — Department of Metabolism, Digestion and Reproduction, Imperial College London
Locations (3):
- United Kingdom (3):
  - Royal Marsden NHS Foundation Trust (Chelsea), London
  - Imperial College NHS Foundation Trust, Charing Cross Hospital, London
  - The Royal Marsden NHS Foundation Trust (Sutton), Sutton

IPD SHARING:
Plan to Share IPD: Yes
Final versions of the anonymised databases and data files will be made available to the wider research community including other groups interested in breast cancer margin technologies and clinical applications / translation of mass spectroscopy.
  Imperial College London retains copyright of the databases and data files. As part of the registration process users must agree to the conditions in the Data User Agreement including: restrictions against attempting to identify participants; destruction of data after analysis; reporting responsibilities (i.e. any publication arising as a result of sharing of the data will need to acknowledge the project PIs: Zoltan Takats & Daniel Leff and Cancer Research United Kingdom as the funder); respecting the embargo period regarding publication; proper acknowledgment of the data resource and restrictions on sharing with third parties. A Data User Agreement must be signed before access to the data is permitted.
Supporting Information: Study Protocol, ICF
Time Frame: 6 months after study completion
Access Criteria: Researchers will be able to access data upon a written request to the project PIs (Zoltan Takats & Daniel Leff).